CLINICAL TRIAL: NCT07265648
Title: Characterization, Perceived Stress Scores, Nut Consumption and Bowel Patterns of a Healthy Adult Population in Northern California: A Pilot Study
Brief Title: Assessing Diet, Stress Scores, and Other Health Metrics in Healthy Northern California Adults
Status: Completed | Type: Observational
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2337131
Record Dates: First submitted 2025-11-20; First posted 2025-12-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Stress; Stool Frequency; Food Allergies; Diet Surveys; Demographic Data
Keywords: Survey; Observational Study; Online Survey; Stress; Diet; allergens
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults living in and around Davis, CA: Adults 18-65 years old, currently living in Yolo, Sacramento, Solano, Sutter, or Placer counties
  Interventions: Other: Online Survey

INTERVENTIONS:
Other: Online Survey — Online survey containing a Perceived Stress Score - 4 instrument, a modified food frequency questionnaire, and will measure reported age, sex, geographical location, usage of prescription medications, food allergies, and stool frequency and consistency.

SUMMARY:
The purpose of this study is to gather health and nutrition data from the population of Davis, CA and surrounding areas. This data will be used to help us test and improve our study procedures for a larger planned study on peanut consumption and effects on cardiovascular disease (CVD) risk.

DETAILED DESCRIPTION:
Participants will be recruited to complete an online survey asking questions about their stress levels, nut consumption, bowel patterns, body measurements, and county of residence. This data will be used to gain insight into the characteristics of this population.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years old
* Currently living in Yolo, Sacramento, Solano, Sutter, or Placer counties
* Able to complete an online survey written in English, on mobile phone, tablet, or computer

Exclusion Criteria:

* Previous participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18-65 years old, currently living in Yolo, Sacramento, Solano, Sutter, or Placer counties
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2025-12-08 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Score | Baseline
  Measured using a validated tool for assessing perceived psychosocial stress within the last month, the Perceived Stress Scale 4 (PSS-4). Participants will report their answers to 4 questions in frequencies ranging from "Never" to "Very Often" on a 5 point scale
Nut Consumption Frequency and Quantity | Baseline
  Participants will input frequencies of nut and nut butter consumption and amounts of nuts and nut butter consumed in a typical month, using a modified food frequency questionnaire. Frequency will be reported as values ranging from "Never" to "6 or more times a week". Nut and nut butter consumption will be reported in cups and tablespoons

SECONDARY OUTCOMES:
Consumption Frequency of Nut-Containing Foods | Baseline
  Reported as monthly consumption of nut containing foods (granola, cereal, pastries, breads, or other snacks or sweets) in frequencies ranging from "Never" to "6 or more times per week"
Prevalence of Food Allergies | Baseline
  Reported as allergies to any of 9 common food allergens: (Peanuts, Tree Nuts, Egg, Wheat, Soy, Shellfish, Fish, Sesame, and Milk)
Stool Frequency | Baseline
  Reported as usual number of bowel movements per week
Stool Consistency | Baseline
  Reported using images of Bristol Scale stool types
Body Mass Index (BMI) | Baseline
  Calculated using participant-reported height and weight
Prescription Drug Use | Baseline
  Participants will confirm or deny intake of medications from 6 categories: (Asthma medications, Antibiotics or antivirals, weight loss medications, cholesterol or lipid lowering medications, blood pressure medications, or psychiatric medications)
Age | Baseline
  Reported as age in years
Biological Sex | Baseline
  Reported as sex assigned at birth
Geographic Data | Baseline
  Reported as current county of residence

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Snodgrass, PhD, Principal Investigator — United States Department of Agriculture - Western Human Nutrition Research Center
Locations (1):
- USDA Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No